CLINICAL TRIAL: NCT02027974
Title: ICONACY Hip Clinical Data Acquisition (13-1-M-239)
Brief Title: Post-Market Study of the ICONACY Hip System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Iconacy Orthopedic Implants, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1-M-239
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Joint Disease
Keywords: Hip; Arthroplasty; Arthroplasties; Prosthesis; Iconacy; Osteoarthritis; Arthritis; THA; THR; DJD
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iconacy Hip System (Active Comparator): Iconacy hip system prosthesis components
  Interventions: Device: Iconacy Hip System
- Stryker Accolade Hip System (Active Comparator): Stryker Accolade hip system prosthesis components
  Interventions: Device: Stryker Accolade Hip System

INTERVENTIONS:
Device: Iconacy Hip System — Comparison of Iconacy I-Hip system to the Stryker Accolade hip system using a randomized study.
  Other Names: Iconacy I-Hip; I-Hip; iHip
  Arms: Iconacy Hip System
Device: Stryker Accolade Hip System — Comparison of Iconacy I-Hip system to the Stryker Accolade hip system using a randomized study.
  Other Names: Accolade
  Arms: Stryker Accolade Hip System

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the Iconacy Hip System for total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* This must be a primary hip replacement on this hip
* Patient is 30 years of age or older
* Have hip joint disease related to one or more of the following: degenerative joint disease, including osteoarthritis or traumatic arthritis
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures

Exclusion Criteria:

* Is younger than 30 years of age
* If there has been a total hip replacement on this hip in the past (no revisions allowed in study)
* Infection, or history of infection, acute or chronic, local or systemic
* Alcoholism or other addictions
* Muscular, neurological or vascular deficiencies which compromise the affected extremity
* Obesity(BMI>45)
* Insufficient bone quality
* Loss of ligamentous structures
* High levels of physical activity
* Materials sensitivity
* Prisoner
* Mental conditions that may interfere with the patient's ability to give an informed consent or willingness to fulfill the study requirements
* Patient is pregnant
* Is not able to read English language

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic success | 2 years
Harris Hip Score must be > or = 80 at 2 years | 2 years
Oxford Hip Score > 40 points at 2 years | 2 years

SECONDARY OUTCOMES:
Patient Satisfaction at 1, 2, and 3 years | 1, 2, and 3 years
Improvement in Harris Hip Score from pre-surgery to 1, 2, and 3 years | 1, 2, and 3 years
Improvements in Oxford Hip Score from pre-survey to 1, 2, and 3 years | 1, 2, and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: William A Hodge, MD, Principal Investigator — Eastern Maine Medical Center